CLINICAL TRIAL: NCT07173413
Title: Evaluating the Quality of Telephone Follow-Up After Spine Surgery: A Non-Inferiority Study
Brief Title: Assessing the Quality of Telephone Follow-Up After Spine Surgery
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Jacob Christiansen Gandløse, Principle investigator, Aalborg University Hospital
Other Study IDs: K2025-124
Record Dates: First submitted 2025-08-27; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
Keywords: low back pain; surgery
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing surgery for low back pain receiving in-person physiotherapy follow-up: Patients undergoing surgery for low back pain receiving in-person physiotherapy follow-up
  Interventions: Other: In person post-operative physiotherapy follow-up
- Patients undergoing surgery for low back pain receiving telephone physiotherapy follow-up: Patients undergoing surgery for low back pain receiving telephone physiotherapy follow-up
  Interventions: Other: Telephone post-surgery physiotherapy follow-up

INTERVENTIONS:
Other: Telephone post-surgery physiotherapy follow-up — Post-operative physiotherapy follow-up delivered via a structured telephone consultation. The session focuses on recovery after lumbar spine surgery, addressing pain management, mobility, exercise recommendations, and guidance on daily activities. The physiotherapist evaluates the patient's status verbally, answers questions, and provides tailored advice to support safe rehabilitation without requiring the patient to attend the hospital physically.
  Other Names: Telephone physiotherapy follow-up
  Groups: Patients undergoing surgery for low back pain receiving telephone physiotherapy follow-up
Other: In person post-operative physiotherapy follow-up — Post-operative physiotherapy follow-up delivered as an in-person consultation at the hospital. The session includes assessment of recovery after lumbar spine surgery, hands-on evaluation if needed, and tailored advice on pain management, mobility, exercise progression, and daily activity. This format allows the physiotherapist to physically observe and, if relevant, demonstrate exercises to ensure correct performance and safe rehabilitation.
  Groups: Patients undergoing surgery for low back pain receiving in-person physiotherapy follow-up

SUMMARY:
The aim of this study is to investigate whether the quality of physiotherapy follow-up after spinal surgery can be maintained when conducted by telephone rather than in-person. The study is motivated by the desire to save healthcare resources and reduce the environmental impact of patient travel. Data from patient records, including age, sex, surgery procedure, use of pain medication, and time spent on either phone or in-person follow-ups, will be collected to evaluate whether telephone-based follow-up is an effective and sustainable alternative for post-operative care.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness and patient experience of telephone-based versus in-person physiotherapy follow-up after spinal surgery. Patients are allocated to one of two groups based on the day of the week they undergo surgery. This allocation determines whether the patient receives a follow-up assessment by telephone or in-person with a physiotherapist.

Following their assigned follow-up, patients are asked to complete questionnaires via REDCap regarding their satisfaction with the follow-up, regardless of the modality. These questionnaires also collect information on pain, physical function, and health-related quality of life. In addition to the initial assessment immediately after the follow-up, patients are sent the same questionnaires again at one and three months post-surgery.

The primary objective of the study is to compare outcomes between the two groups, evaluating whether telephone-based follow-up provides a comparable level of satisfaction, pain management, functional recovery, and quality of life to traditional in-person follow-up. The results will inform whether telephone follow-up is a viable and resource-efficient alternative to in-person assessments while maintaining high standards of post-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone lumbar spine surgery at the Department of Neurosurgery, Aalborg University Hospital, Aalborg, Denmark.
* Able to read and understand Danish.

Exclusion Criteria:

* Withdrawel of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing lumbar spine surgery at Aalborg University Hospital, Neurosurgical Department, who are able to read and understand Danish and consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | Immediately after the postoperative follow-up consultation with the physiotherapist, 1 month, and 3 months post-surgery.
  The ODI is a validated questionnaire assessing disability related to low back pain. It includes 10 items covering pain and daily functional limitations. Each item is scored from 0 to 5, where 0 represents minimal limitation and 5 represents severe limitation. The total score ranges from 0 to 50, with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Health related quality of life | Immediately after the postoperative follow-up consultation with the physiotherapist, 1 month, and 3 months post-surgery.
  The EQ-5D-5L questionnaire is a standardized measure of health-related quality of life recommended for multimorbidity research. The EQ-5D-5L assesses health status across five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-point ordinal scale ranging from 1 (indicating no problems) to 5 (indicating extreme difficulties) The EQ-5D index score can be regarded as a continuous outcome and ranges from -0.624 to 1, with higher scores indicating better general health and quality of life.
Patient Satisfaction with Follow-up (Modified CSQ-8) | Immediately after the postoperative follow-up consultation with the physiotherapist, 1 month, and 3 months post-surgery.
  Patient satisfaction will be assessed using a modified version of the validated Client Satisfaction Questionnaire-8 (CSQ-8). The original 8-item instrument measures overall satisfaction with healthcare services. For this study, the questionnaire has been adapted to specifically reflect the follow-up consultation with the physiotherapist, ensuring that responses relate to the guidance and instruction provided during the post-operative follow-up. Modifications include context-specific wording, such as "...based on the follow-up consultation with the physiotherapist," while maintaining the original structure and response options. Higher scores indicate greater satisfaction.
Back and leg pain (VAS, 0-100 mm) | Immediately after the postoperative follow-up consultation with the physiotherapist, 1 month, and 3 months post-surgery.
  Leg pain and back pain will be assessed using a 0-100 mm Visual Analog Scale (VAS), where 0 represents "no pain" and 100 represents "worst imaginable pain."

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Aalborg University Hospital, Aalborg, Denmark., Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including questionnaire responses, pain scores, and functional outcomes) will be made available upon reasonable request to qualified researchers. Data will be shared after publication of the main study results. Requests must include a research proposal and be approved by the study investigators. Data will be shared under a data use agreement to ensure confidentiality and compliance with Danish data protection regulations.